CLINICAL TRIAL: NCT04363229
Title: Psychological Impact of COVID19 Among Doctors in Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Roshdy Elkhayat, lecturer of public health, Assiut University
Other Study IDs: pshycological impact COVID19
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Occupational Stress
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: maslach burnout inventory questionnair — The Maslach Burnout Inventory (MBI) is an introspective psychological inventory consisting of 22 items pertaining to occupational burnout
  Other Names: GHQ-12 questionnair

SUMMARY:
study aimed to investigate the psychological impact of corona virus among doctor in Assiut University Hospitals, mainly stress and burn out will be assessed

DETAILED DESCRIPTION:
Prolonged exposure to stressful working environments resulting in a state of physical and emotional depletion and burnout. Nowadays, while facing corona virus, health care workers are on the front line and directly assist in diagnosis, caring and treatment of patients with COVID, thus keeping them at higher risk developing psychological distress and other mental health symptoms.

According to previous studies, during the outbreaks of severe acute respiratory syndrome (SARS) and Middle East respiratory syndrome (MERS), frontline medical staff had reported high levels of stress that resulted in posttraumatic stress disorder (PTSD)

A lot of factors contribute to increase mental effect among healthcare workers as increasing the suspected cases and workload , depletion of personal protective equipment's , drug shortage and feeling inadequately supported .

In Toronto study(2008), four major risk factors for stress among medical staff during the SARS outbreak were identified; including the perception of the medical of their risk of infection, the impact of SARS on their work, feelings of depression, and working in high-risk medical units. moreover, there are other factors as social stigmatization and contact with infected patients, also has previously been shown to be associated with increased levels of stress and anxiety in medical staff .

ELIGIBILITY:
Inclusion Criteria:

* all doctors currently working in assiut University hospitals

Exclusion Criteria:

* no exclusion critiria

Min Age: 22 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Doctors currently working in Assiut University Hospitals in all titles: resident doctors, assistant lecturer, lecturer, assistant professor and professor
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
The MBI-HSS (MP) addresses three scales:Emotional Exhaustion ,Depersonalization and Personal Accomplishment | baseline
  Emotional Exhaustion measures feelings of being emotionally overextended and exhausted by one's work.
  Depersonalization measures an unfeeling and impersonal response toward patients.
  Personal Accomplishment measures feelings of competence and successful achievement in one's work.
  All MBI items are scored using a 7 level frequency scale from "never" to "daily." Initial development had 3 components: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout

SECONDARY OUTCOMES:
GHQ-12 questionnaire for measuring of current mental health | baseline
  The scale asks whether the respondent has experienced a particular symptom or behavior recently. Each item is rated on a four-point scale (less than usual, no more than usual, rather more than usual, or much more than usual); and for example when using the GHQ-12 it gives a total score of 36 or 12 based on the selected scoring methods.
  it measure social dysfunction, anxiety and depression and loss of confidence

REFERENCES:
- See also: Psychological Impact and Coping Strategies of Frontline Medical Staff in Hunan Between January and March 2020 During the Outbreak of Coronavirus Disease 2019 (COVID-19) in Hubei, China — https://www.ncbi.nlm.nih.gov/research/coronavirus/publication/32291383
- See also: The emotional impact of Coronavirus 2019-nCoV (newCoronavirusdisease) — https://www.ncbi.nlm.nih.gov/pubmed/32199182